CLINICAL TRIAL: NCT05802732
Title: Diagnostic Accuracy Of Stool Antigen In Diagnosis Of Helicobacter Pylori Infection In Children
Brief Title: Stool Antigen In Diagnosis Of Helicobacter Pylori
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yosra Alaa Abd El-baset Ali Khallaf, Principal Investigator, Assiut University
Other Study IDs: DAOSADOHPIC
Record Dates: First submitted 2023-03-25; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Stool Antigen test — Correlation between the result of endoscopic biopsy and stool antigen test

SUMMARY:
Helicobacter pylori is among the most common bacterial infections in humans. Helicobacter pylori is a Gram-negative, S -shaped rod .The most likely mode of transmission is fecal-oral or oral-oral. Helicobacter pylori infection is acquired in early life and continues to have a high prevalence, especially in developing countries. Growing antibiotic-resistant strains necessitate adapted treatments. The majority of children with Helicobacter pylori infection remain asymptomatic, although a percentage of the infected children do develop Helicobacter. pylori-associated diseases. Helicobacter pylori is closely associated with the development of gastritis, gastric or duodenal ulcers. Helicobacter pylori infection can manifest with abdominal pain or vomiting and, less often, refractory iron deficiency anemia or growth retardation. Helicobacter pylori can be associated, though rarely, with chronic autoimmune thrombocytopenia. Anemia, idiopathic thrombocytopenic purpura, short stature, and sudden infant death syndrome (SIDS) have also been reported as possible extra-gastric manifestations of Helicobacter pylori infection . The diagnosis of Helicobacter pylori infection is made histologically by demonstrating the organism in the biopsy specimens. 13 C-urea breath tests and stool antigen tests are reliable noninvasive methods of detecting Helicobacter pylori infection in patients who do not require endoscopic evaluation. However, some guidelines recommend that non-invasive assessment methods are reserved to determine whether Helicobacter pylori has been eradicated not for diagnosis .However Helicobacter pylori-associated gastritis may, however, be an incidental histopathologic finding during upper endoscopy performed for unrelated indications such as the diagnosis of inflammatory bowel disease, or celiac disease.

ELIGIBILITY:
Inclusion Criteria:

- 1. Children and adolescents between 4 and 18 years old having chronic or reccurent unexplained dyspeptic symptoms (epigastric pain, post prandial fullness, early satiety, bleching, heart burn, bloating, flatulence, regurgitation, nausea, vomiting and/ or halitosis)(Miwa et al.,2012) and/ or non variceal hematemesis

2. The dyspeptic symptoms should be present at least 2months duration , which doesn't need to be consecutive, during the previous 6 months.(Rasquin et al., 2006)

Exclusion Criteria:

- 1. Patients who received anti sectertory drugs and/ or antibiotics in the previous 4 weeks before endoscopy.

2. Patients less than 4years and more than 18 years old.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include children and adolescents recruited from the Gastroenterology, Hepatology And Endoscopy Unit at Assuit University, Children's Hospital.
Sampling Method: Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
detect the diagnostic accuracy of stool Ag test in diagnosis of H.pylori infction in children and adolescents | over one year
  Patients presented with chronic or recurrent unexplained dyspeptic symptoms and/or non variceal hematemesis will be submitted for stool antigen test

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moubri M, Kalach N, Larras R, Berrah H, Mouffok F, Guechi Z, Cadranel S. Adapted first-line treatment of Helicobacter pylori infection in Algerian children. Ann Gastroenterol. 2019 Jan-Feb;32(1):60-66. doi: 10.20524/aog.2018.0317. Epub 2018 Oct 3. PMID 30598593
- [Background] Kato S, Shimizu T, Toyoda S, Gold BD, Ida S, Ishige T, Fujimura S, Kamiya S, Konno M, Kuwabara K, Ushijima K, Yoshimura N, Nakayama Y; Japanese Society for Pediatric Gastroenterology, Hepatology and Nutrition. The updated JSPGHAN guidelines for the management of Helicobacter pylori infection in childhood. Pediatr Int. 2020 Dec;62(12):1315-1331. doi: 10.1111/ped.14388. PMID 32657507
- [Background] Galicia Poblet G, Alarcon Cavero T, Alonso Perez N, Borrell Martinez B, Botija Arcos G, Cilleruelo Pascual ML, Gonzalez Martin LM, Hernandez Hernandez A, Martinez Escribano B, Ortola Castells X, Rizo Pascual J, Urruzuno Telleria P, Vegas Alvarez AM. Management of Helicobacter pylori infection in the pediatric age. An Pediatr (Engl Ed). 2021 Nov;95(5):383.e1-383.e9. doi: 10.1016/j.anpede.2021.05.004. Epub 2021 Oct 9. PMID 34642127
- [Background] Jones NL, Koletzko S, Goodman K, Bontems P, Cadranel S, Casswall T, Czinn S, Gold BD, Guarner J, Elitsur Y, Homan M, Kalach N, Kori M, Madrazo A, Megraud F, Papadopoulou A, Rowland M; ESPGHAN, NASPGHAN. Joint ESPGHAN/NASPGHAN Guidelines for the Management of Helicobacter pylori in Children and Adolescents (Update 2016). J Pediatr Gastroenterol Nutr. 2017 Jun;64(6):991-1003. doi: 10.1097/MPG.0000000000001594. PMID 28541262
- [Background] Huh CW, Kim BW. [Diagnosis of Helicobacter pylori Infection]. Korean J Gastroenterol. 2018 Nov 25;72(5):229-236. doi: 10.4166/kjg.2018.72.5.229. Korean. PMID 30642138
- [Background] Breckan RK, Paulssen EJ, Asfeldt AM, Kvamme JM, Straume B, Florholmen J. The All-Age Prevalence of Helicobacter pylori Infection and Potential Transmission Routes. A Population-Based Study. Helicobacter. 2016 Dec;21(6):586-595. doi: 10.1111/hel.12316. Epub 2016 May 12. PMID 27172105
- [Background] Qualia CM, Katzman PJ, Brown MR, Kooros K. A report of two children with Helicobacter heilmannii gastritis and review of the literature. Pediatr Dev Pathol. 2007 Sep-Oct;10(5):391-4. doi: 10.2350/06-09-0159.1. PMID 17929990
- [Background] Rasquin A, Di Lorenzo C, Forbes D, Guiraldes E, Hyams JS, Staiano A, Walker LS. Childhood functional gastrointestinal disorders: child/adolescent. Gastroenterology. 2006 Apr;130(5):1527-37. doi: 10.1053/j.gastro.2005.08.063. PMID 16678566
- [Background] Miwa H, Ghoshal UC, Gonlachanvit S, Gwee KA, Ang TL, Chang FY, Fock KM, Hongo M, Hou X, Kachintorn U, Ke M, Lai KH, Lee KJ, Lu CL, Mahadeva S, Miura S, Park H, Rhee PL, Sugano K, Vilaichone RK, Wong BC, Bak YT. Asian consensus report on functional dyspepsia. J Neurogastroenterol Motil. 2012 Apr;18(2):150-68. doi: 10.5056/jnm.2012.18.2.150. Epub 2012 Apr 9. PMID 22523724